CLINICAL TRIAL: NCT06055985
Title: A Multicenter Phase 2, Double-blind, Placebo-controlled, Randomized, Parallel-group Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of UCB0022 in Study Participants With Advanced Parkinson's Disease
Brief Title: A Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of UCB0022 in Study Participants With Advanced Parkinson's Disease
Acronym: ATLANTIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PD0060
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Phase 2; UCB0022; wearing-off; motor fluctuations
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor and CRO staff is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- UCB0022-Dose A (Experimental): Study participants randomized to this arm will receive UCB0022 Dose A orally administered as tablet during the Treatment Period.
  Interventions: Drug: UCB0022
- UCB0022-Dose B (Experimental): Study participants randomized to this arm will receive UCB0022 Dose B orally administered as tablet during the Treatment Period.
  Interventions: Drug: UCB0022
- Placebo (Placebo Comparator): Study participants randomized to this arm will receive matching placebo orally administered as tablet during the Treatment Period.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Study participants will receive placebo orally administered as tablet at pre-specified time points during the study.
  Arms: Placebo
Drug: UCB0022 — Study participants will receive UCB0022 dose A or B orally administered as tablet at pre-specified time points during the Treatment Period.
  Arms: UCB0022-Dose A; UCB0022-Dose B

SUMMARY:
The primary purpose of this study is to demonstrate the superiority of UCB0022 as an adjunctive treatment to stable dose of standard-of-care (SoC) (including at least levodopa therapy) over placebo with regard to motor fluctuations time spent in the OFF state (OFF time) in study participants with advanced Parkinson's Disease (PD).

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be 35 to 85 years of age (inclusive) at the time of signing the informed consent form (ICF)
* Study participant is diagnosed with Parkinson's disease (PD) (based on the United Kingdom Parkinson's Disease Society Brain Bank Diagnostic criteria performed at the Screening Visit) and diagnosed ≥5 years before the Screening Visit (based on historical medical- information documented by the investigator)
* Study participant has significant daily motor fluctuations
* Study participant is able to complete a Hauser PD symptoms diary and differentiate between the ON and OFF states
* Study participant is responsive to levodopa and currently receiving treatment with oral daily doses of levodopa combination (levodopa/carbidopa or levodopa/benserazide) with or without oral adjunctive antiparkinsonian therapies (based on historical clinical data)
* Study participant has disease severity Stages I-III (modified Hoehn and Yahr staging) during ON state
* Study participant agrees to not post personal medical data or information related to the study on social media until study completion
* Study participant has body weight ≥45 kg and body mass index within 18 to 30 kg/m^2 (inclusive)
* Study participant may be male or female:

  1. A male study participant must agree to use contraception during the Treatment Period and for at least 2 weeks after the last dose of study treatment and refrain from donating sperm during this period
  2. A female study participant must not be a woman of childbearing potential (WOCBP)

Exclusion Criteria:

* Study participant is diagnosed with any form of Parkinsonism other than idiopathic PD (eg, atypical or secondary Parkinsonism)
* Study participant is diagnosed with dementia or has important cognitive dysfunction, as determined by Montreal Cognitive Assessment (MoCA) <23 at screening
* Study participant has a history of neurosurgical intervention for PD (including DBS, thalamotomy, and experimental cell therapy or gene therapy)
* Participant has a severe peak dose or biphasic dyskinesia at screening, defined by Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) items 4.2 score 4 or as per investigator opinion
* Participant has a history of major depression or psychotic disorder or any other psychiatric condition within the past 5 years, that, as per investigator opinion, could jeopardize or would compromise the study participant's ability to participate in the study
* Study participant has a history of narrow angle glaucoma
* Study participant has a history of melanoma
* Study participant has current untreated hypertension
* Study participant has a history of hypertensive crisis and/or hypertensive encephalopathy, unless the underlying cause was unequivocally identified and has been removed
* Study participant has orthostatic hypotension requiring medication or a current history of "clinically significant" orthostatic hypotension as per the investigator's opinion (eg, recurrent orthostatic presyncope or syncope)
* Study participant has a history over the past 12 months or between the Screening and Baseline Visits of any clinically significant arrythmia, myocardial infarction, stroke, transient ischemic attack, moderate or severe congestive heart failure (either New York Heart Association Class III or IV or known ejection fraction <40%)

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Visit 9 (Day 70) in the average number of hours/day of OFF time, as assessed by the study participant-completed Hauser PD symptoms diary over 3 consecutive days | From Baseline (Day 1) to Visit 9 (Day 70)
  The Hauser Parkinson's disease (PD) symptoms diary is a study participant-completed diary that records the daily ON time and OFF time of study participants with PD with motor fluctuations and dyskinesia.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From Baseline (Day 1) to End of Safety Follow-up (up to Week 12)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP. TEAEs are defined as AEs starting after the time of first IMP administration up to and including 2 weeks after the final dose.
Incidence of treatment-emergent serious adverse events (SAEs) | From Baseline (Day 1) to End of Safety Follow-up (up to Week 12)
  A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent disability/incapacity
  * Is a congenital anomaly/birth defect
  * Important medical events Treatment-emergent AEs are defined as those AEs that have a start date on or following the first dose of investigational medicinal product (IMP).
Incidence of TEAEs leading to withdrawal from the study | From Baseline (Day 1) to End of Safety Follow-up (up to Week 12)
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of IMP, whether or not considered related to the IMP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP. TEAEs are defined as AEs starting after the time of first IMP administration up to and including 2 weeks after the final dose.
Average Ctrough of UCB0022 and its active N-desmethyl-UCB0022 metabolite at Visit 9 (Day 70) | at Visit 9 (Day 70)
  Ctrough: The predose observed plasma concentration (average, per visit) will be plotted and depicted graphically to assess trajectory to steady-state for parent and active metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (61):
- United States (61):
  - Pd0060 50506, Phoenix, Arizona
  - Pd0060 50590, Scottsdale, Arizona
  - Pd0060 50608, Little Rock, Arkansas
  - Pd0060 50519, Fountain Valley, California
  - Pd0060 50428, Fresno, California
  - Pd0060 50601, Loma Linda, California
  - Pd0060 50589, Los Alamitos, California
  - Pd0060 50587, Los Angeles, California
  - Pd0060 50452, Pasadena, California
  - Pd0060 50598, Englewood, Colorado
  - Pd0060 50628, New Haven, Connecticut
  - Pd0060 50610, Newark, Delaware
  - Pd0060 50600, Altamonte Springs, Florida
  - Pd0060 50616, Aventura, Florida
  - Pd0060 50596, Boca Raton, Florida
  - Pd0060 50524, Bradenton, Florida
  - Pd0060 50647, DeLand, Florida
  - Pd0060 50577, Doral, Florida
  - Pd0060 50584, Hollywood, Florida
  - Pd0060 50582, Miami, Florida
  - Pd0060 50579, Miami, Florida
  - Pd0060 50449, Miami, Florida
  - Pd0060 50580, Miami, Florida
  - Pd0060 50597, Naples, Florida
  - Pd0060 50591, Ocala, Florida
  - Pd0060 50605, Port Orange, Florida
  - Pd0060 50620, St. Petersburg, Florida
  - Pd0060 50603, Tampa, Florida
  - Pd0060 50585, Winter Park, Florida
  - Pd0060 50075, Augusta, Georgia
  - Pd0060 50595, Indianapolis, Indiana
  - Pd0060 50319, Iowa City, Iowa
  - Pd0060 50074, Kansas City, Kansas
  - Pd0060 50561, Lexington, Kentucky
  - Pd0060 50615, Boston, Massachusetts
  - Pd0060 50085, Boston, Massachusetts
  - Pd0060 50627, North Dartmouth, Massachusetts
  - Pd0060 50110, Ann Arbor, Michigan
  - Pd0060 50545, East Lansing, Michigan
  - Pd0060 50386, Farmington Hills, Michigan
  - Pd0060 50613, Grand Rapids, Michigan
  - Pd0060 50614, New York, New York
  - Pd0060 50521, New York, New York
  - Pd0060 50612, Raleigh, North Carolina
  - Pd0060 50087, Centerville, Ohio
  - Pd0060 50622, Cleveland, Ohio
  - Pd0060 50076, Columbus, Ohio
  - Pd0060 50604, Dayton, Ohio
  - Pd0060 50527, Toledo, Ohio
  - Pd0060 50398, Tulsa, Oklahoma
  - Pd0060 50607, Portland, Oregon
  - Pd0060 50619, Rock Hill, South Carolina
  - Pd0060 50496, Round Rock, Texas
  - Pd0060 50568, San Antonio, Texas
  - Pd0060 50537, Salt Lake City, Utah
  - Pd0060 50143, Henrico, Virginia
  - Pd0060 50534, Virginia Beach, Virginia
  - Pd0060 50440, Bellevue, Washington
  - Pd0060 50292, Kirkland, Washington
  - Pd0060 50419, Spokane, Washington
  - Pd0060 50402, Crab Orchard, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if a determination is made that the data cannot be adequately anonymized.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal
URL: http://vivli.org